CLINICAL TRIAL: NCT04851808
Title: Estimating the Burden of Chronic Respiratory Diseases (CRD) in Bangladesh Using the 4 Country Chronic Respiratory (4CCORD) Study Tools
Brief Title: Chronic Respiratory Disease Burden in Bangladesh
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Child Health Research Foundation, Bangladesh (Other)
Collaborators: University of Edinburgh (Other); KEM Hospital Research Centre (Other)
Responsible Party: Sponsor
Other Study IDs: CHRF002
Record Dates: First submitted 2021-04-15; First posted 2021-04-20 (Actual); Last update posted 2021-04-20 (Actual); Status verified 2021-04

CONDITIONS: Chronic Respiratory Disease; COPD
Keywords: Chronic Respiratory Disease; Spirometry; COPD Surveillance; Developing Countries
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Chronic Respiratory Disease (CRD), particularly asthma and chronic obstructive pulmonary disorders (COPD) are leading causes of mortality and reduced quality of life due to its wide-reported association with other multi-morbidities.There is limited knowledge on the burden of CRD in the rural communities in Bangladesh due to poor awareness on the impact of CRD on quality of life and unavailability of diagnostic facilities due to weaker primary healthcare settings. The study aims to estimate the CRD burden in Bangladesh in a large representative population to draw the attention of policy makers to the creation of social awareness and improvement of primary healthcare infrastructure for respiratory disease in Bangladesh.

The study is a prospective observational one in nature. The study will be implemented in Mirzapur, a rural sub-district of Tangail district in Bangladesh within the period of February to May 2021. A total of 981 participants will be enrolled from the study. Verbal consent will be taken initially. Participants who are assessed to be COVID-19 negative will be invited for a visit to the mobile clinic following national health guidelines to perform the spirometry. The study team will provide an information sheet (written in local language) that describes the study aim and objectives with potential risk benefits to the participants. All participants will be enrolled through written consent and satisfactory response to the patient information sheet.

The Research Assistant (RA) will collect the relevant metadata such as demographics, information on risk factors, screening questionnaires relevant to asthma and COPD, reported health status and symptoms related to CRD etc. from the participant after obtaining the written consent. Data quality will be ensured by the Field Research Supervisor through checking all the collected information. The enrolled participants will undergo spirometry for the evaluation of their lung function. Spirometry will be collected by trained personnel and will be quality checked by an expert panel at CHRF. Repeated collection will take place in the event if the test results do not pass quality checking. Participant will also be invited to the study clinic within the next 10 days after assessment for any further clinical assessment that is deemed necessary by the study physician. The collected data and spirometry reports will be reviewed to evaluate the CRD patient in terms of their disease. The study will analyse the rate of CRD burden stratified by age, sex, and income group. The productivity loss will be measured in terms of work hours lost due to CRDs.

DETAILED DESCRIPTION:
BACKGROUND Chronic respiratory diseases (CRD), particularly asthma and chronic obstructive pulmonary disease (COPD) are leading causes of mortality and associated with multi-morbidity, leading to reduced productivity worldwide[1, 2]. We have limited data on the prevalence of CRD in Bangladesh, especially from the rural communities, where poor awareness and care-seeking behaviour, is compounded by the unavailability of diagnostic facilities and presence of weak primary health infrastructures. Determining the burden of CRD in these settings is thus challenging.

The RESPIRE 4-Country Chronic Respiratory Disease (4CCORD) pilot study, revealed a high prevalence of asthma (7%) and COPD (8%) in Bangladesh including many who were unaware of having mild airway obstruction and thus susceptible to CRD in future (unpublished data). Early diagnosis of these diseases could facilitate better primary prevention (abstaining from the exposure to harmful risk factors) and management to prevent deterioration.

The 4CCORD study aimed to validate the research tools and methodologies to detect the CRD cases at the community level. This study collected information from only 100 participants, thus lacked power drawing inference on the burden of CRD in the Bangladeshi population. With the support of RESPIRE and utilising the Child Health Research Foundation (CHRF) existing infrastructure, we want to survey an adequate sample to estimate the CRD burden in Bangladesh confidently. These data will help to draw the attention of the policymakers to these important diseases and create social awareness of CRD in Bangladesh.

STUDY AIM and OBJECTIVES To reduce the mortality and morbidity associated with CRD in Bangladesh by providing data on the health and economic burden of these diseases.

OBJECTIVES PRIMARY OBJECTIVE

1. To estimate the prevalence of CRD at the community level in Bangladesh using the screening questionnaire and objective measurements
2. To determine the risk factors for CRD in the community settings in Bangladesh SECONDARY OBJECTIVES

a. To determine the burden of early-stage asthma and COPD in the community settings in Bangladesh b. To assess the loss of productivity and impact on the quality of life due to CRD in Bangladesh c. To determine the healthcare-associated costs with CRD in community settings in Bangladesh

STUDY DESIGN This is a prospective observational study. This study protocol will be implemented from January 2021 to April 2021. The participants will be recruited from Mirzapur, a rural Upazila (sub-district) of Tangail district in Bangladesh; located 65 km north of Dhaka. A list of eligible study participants (currently residing in the study area and are above 18 years of age) will be generated from the existing demographic surveillance system (DSS) database. The eligible participants will be reached over telephone by a research assistant to inform the study objectives and procedures. Those who provides verbal consent will be asked i) whether the participants or any household member been diagnosed with COVID-19/coronavirus disease in the past 14 days, ii) currently any of the household member have COVID-19 sign/symptoms (dry cough, shortness of breath or difficulty breathing, fever or chills, sore throat, loss of taste or smell, vomiting or diarrhoea), and iii) Whether any household member currently under quarantine or in self-isolation due to contact with a case of COVID-19/coronavirus disease or because of an order by a physician or public health authority?. Participants who provide negative answer of all three questions mentioned above will be asked to attend a mobile clinic to perform the spirometry. Only three participants will be asked to attend a session to minimise the risk of COVID-19 infection. The participants will be seated in a waiting room maintaining social distance and askinvited for the interview in an isolatedprivate room one by one.

The mobile team, consist a research assistant, a field supervisor and a medical technologist/nurses will perform the spirometry at an open place following the national health guidelines. Research assistants (RA) will provide the patient information sheet of the study to the participants and will give satisfactorily answers to the questions raised by the participants. Only participants who provide written consent for their participation in the study will be enrolled in the study. Once the participants provide the consent, RA will collect all the metadata such as demographics, risk factor information, reported heath status etc. from the study participant. A Field Research Supervisor (FRS) will check all information collected by the RA to ensure the data quality..

Each study participant will undergo spirometry to check their lung functions. A nurse/medical technologist will conduct the spirometry tests after receiving appropriate training. All spirometry data will be reviewed by an expert panel at CHRF to ensure the quality of the spirometry. All spirometry data which do not pass the quality will be repeated. Collected data and spirometry reports will be reviewed by a respiratory physician to level the CRD patients and their type of illness. The enrolled participants may be invited to Mirzapur hospital for further clinical examination within the next 10 days of the assessment based on the physician's review and the collected information. The spirometry may be repeated and any other test to be suggested by the physician if needed.

STUDY POPULATION A total number of 981 participants aged more than 18 years will be enrolled in the study.

STUDY PROCEDURES: ASSESSMENTS Screening data collection: After obtaining informed consent from the eligible participants for enrolment, RA will collect the metadata using screening questionnaires (described below) including demographics, risk factors, reported health status from the study participants. Disease burden assessment shall be conducted using COPD Assessment Tool (CAT), GINA Ashtma Control test etc. This will be followed by conducting spirometry using NDD Easyone Air spirometer by trained technologist. The primary spirometry indices will be FEV1, FVC and FEV1/FVC. Spirometry will be performed before and after bronchodilation via two puffs of salbutamol via MDI+spacer. Quality check of the spirometry data generated will be reviewed by the experts on a regular basis and any failure of meeting the quality standards will render repeated collection. Each participant's data will be reviewed by the physicians on a regular basis for assessing CRD based on screening questionnaire and spirometry data. All study team members will be tested periodically (in every 14 days) to ensure that they do not have COVID-19. During the clinical session, they will year protective equipment such as mask, gloves and gown to reduce the exposure risk. All participants will ask to wear mask while not perform the spirometry test. All participants will be ask to seat maintaining social distance. We will provide each participant a sterile flow tube while performing the spirometry. The outside of the spirometer will be cleaned after each session.

Questionnaires: The questionnaires will be comprised of the following section as anticipated:

* Demographic meta-data (age, gender, marital status, occupation)
* Chronic respiratory symptoms (wheeze, cough, chest tightness, shortness of breath) identification, existing respiratory diagnosis, co-morbidities
* Specific screening questionnaire relevant to asthma and/or COPD
* Information on risk factors (smoking habits, fuels used for cooking, types of mosquito repellent used etc)
* Individual burden of disease (e.g. Asthma Control Questionanire, COPD Questionnaire)
* Societal impact (e.g. lost productivity, under-performance)
* Usage of healthcare resources (primary care, secondary care, medication history) A pragmatic balance will be drawn between collecting sufficient detail for as accurate costing as possible while minimising participant burden. The study questionnaires which already used in the 4ccord study will be available both in English and translated into Bengali (local language).

Physician clinical assessment of a random sample: Subsequent clinical examination (see details below) of people diagnosed with CRD and a random sample of screened participants as 'normal' will further confirm the diagnosis achieved by screening. These participants shall be invited to the study clinic/ hospital for further clinical examination within the next 10 days. During the visit, the physician will check the clinical history and perform clinical assessment as necessary. Repeated spirometry and other tests (e.g. Chest X-ray) may be performed at the discretion of the study physician. The physician will confirm participants as asthma and/or COPD and (where possible) the nature of other CRD based on their clinical judgement.

Participants identified with asthma, COPD or other 'CRD' will be advised to seek further advice from their usual clinical services where further investigation can be arranged as per clinical needs. We will request permission to contact their usual clinical advisor for the outcome of any additional test and final conclusion about the diagnosis.

References

1. Braman, S.S., The global burden of asthma. Chest, 2006. 130(1 Suppl): p. 4S-12S.
2. Lopez-Campos, J.L., W. Tan, and J.B. Soriano, Global burden of COPD. Respirology, 2016. 21(1): p. 14-23.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years and above
* Adults residing in the study area with an intention to stay within the auspices of the sites until the completion of the study
* Adults who have consented to take part in the study

Exclusion Criteria:

* Children or adolescents aged less than 18 years
* Adults either outside of the study area or have no intention to stay within the study area
* Adults unable to provide informed consent (e.g. severe cognitive impairment, recent (within one month) myocardial infarction, unstable cardiovascular status, aneurysms (abnormal dilatation of blood vessels), hemoptysis (blood in the cough), pneumothorax (abnormal trapping of air in the walls surrounding the lungs), recent eye, thoracic or abdominal surgery and facial palsy (paralysis of the face muscles))
* Adults unable to complete the study questionnaires in their own language (trained study researchers will be involved to supervise completion and read the questions as necessary )

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult population above the age of 18 residing within the catchment of demographic surveillance system and resident of the Mirzapur upazilla will be taken as sample cohort for this research. The participants will be recruited from Mirzapur, a rural Upazila (sub-district) of Tangail district in Bangladesh; located 65 km north of Dhaka.
Sampling Method: Probability Sample
Enrollment: 981 (Estimated)
Dates: Start 2021-02-01 (Actual); Primary Completion 2021-05-31 (Estimated); Study Completion 2021-09-30 (Estimated)

PRIMARY OUTCOMES:
Chronic Respiratory Diseases | Aged 18 and above at the time of enrollment
  * Wheeze, Cough, Chest tightness and shortness of breath (at least one) present on most days for the last six months OR
  * Respiratory attacks having symptoms lasting than four weeks and occurring at least two times over the last two or more years

SECONDARY OUTCOMES:
Maximum forced expiratory air volume in one second (FEV1) | Aged 18 and above at the time of enrollment
  Lung Function of the Enrolled Participants shall be recorded. Maximum forced expiratory air volume in one second will be reported
Forced Vital Capacity (FVC) | Aged 18 and above at the time of enrollment
  Lung Function of the Enrolled Participants shall be recorded. Forced vital capacity of the lung will be reported
Work Productivity due to Asthma and COPD | Aged 18 and above at the time of enrollment
  The loss of work productivity in hours shall be measured for both Asthma and COPD
Lung Function evaluation through FEV1/FVC ratio | Aged 18 and above at the time of enrollment
  The lung function shall be measured. The ratio of maximum forced expiratory volume in one second (FEV1) and forced vital capacity shall be recorded.
Height of the participant | Aged 18 and above at the time of enrollment
  Height of the participant in meters
Weight of the participant | Aged 18 and above at the time of enrollment
  Weight of the Participant in kg

CONTACTS AND LOCATIONS:
Overall Officials: Aziz Sheikh, BSc, MBBS, MSc, MD, FRCGP,FRCP, Principal Investigator — Usher Institute, University of Edinburgh; Hilary Pinnock, MB, ChB, MRCGP, MD, Study Chair — Usher Institute, University of Edinburgh; Ee M Khoo, MBBS, FBSCH, MRCGP, FAMM, MD, Study Chair — University of Malaya: Kuala Lumpur, Wilayah Persekutuan, MY; Sanjay Juvekar, MSc PhD, Study Chair — KEM University Hospital Pune, India
Locations (1):
- Child Health Research Foundation, Dhaka, Bangladesh

IPD SHARING:
Plan to Share IPD: No
The personal information will be codified and the linkage data will not share with any other organization

REFERENCES:
- [Result] Braman SS. The global burden of asthma. Chest. 2006 Jul;130(1 Suppl):4S-12S. doi: 10.1378/chest.130.1_suppl.4S. PMID 16840363
- [Result] Lopez-Campos JL, Tan W, Soriano JB. Global burden of COPD. Respirology. 2016 Jan;21(1):14-23. doi: 10.1111/resp.12660. Epub 2015 Oct 23. PMID 26494423